CLINICAL TRIAL: NCT00591188
Title: Phase II Study of Capecitabine and Interferon-Alpha in Metastatic Renal Cell Carcinoma Patients With Failure on Interleukin-2 Based Regimens
Brief Title: Capecitabine and Interferon-Alpha in Metastatic Renal Cell Carcinoma Patients With Failure on Interleukin-2 Based Regimens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kidney Cancer Research Bureau (Other)
Responsible Party: Ilya Tsimafeyeu, MD, Kidney Cancer Research Bureau
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRT-003; CRT-003
Record Dates: First submitted 2007-12-28; First posted 2008-01-11 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Carcinoma, Renal Cell
Keywords: kidney cancer, capecitabine, interferon
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Capecitabine; Interferon-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All patients will receive capecitabine and interferon-alpha.
  Interventions: Drug: capecitabine, interferon-alpha

INTERVENTIONS:
Drug: capecitabine, interferon-alpha — Patients who meet inclusion/exclusion criteria will receive combination of study drugs.

SUMMARY:
The aim of this study is to determine preliminary efficacy of capecitabine and interferon-alpha in second-line after interleukin-2 based regimens in patients with MRCC

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed renal carcinoma
* CT-confirmed metastatic sites
* Must have measurable disease, defined as ≥ 1 unidimensionally measurable lesion measured as ≥ 20 mm with conventional techniques OR as ≥ 10 mm with spiral CT scan
* Disease progression after IL-2
* Age 18 or older
* ECOG performance status 1-3
* Life expectancy ≥ 2 months
* WBC ≥ 3,000/mm3
* Platelet count ≥ 100,000/mm3
* Hemoglobin ≥ 7.5 g/dL
* Creatinine ≤ 1.5 mg/dL (2.0 mg/dL in post-nephrectomy patients)
* Total bilirubin ≤ 1.5 mg/dL
* AST ≤ 3.0 times normal
* Alkaline phosphatase ≤ 2.5 times normal (10 times ULN in presence of bone metastases)
* Not pregnant or nursing
* No history of autoimmune
* No history of serious cardiac arrhythmia, congestive heart failure, angina pectoris, or other severe cardiovascular disease (i.e., New York Heart Association class III or IV)
* No CNS metastases by neurologic exam and/or MRI
* No history of seizure disorders
* No local and/or systemic infections requiring antibiotics within 28 days prior to study entry
* No other malignancy
* Written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Evaluate progression-free survival with capecitabine and interferon treatment in metastatic renal cell carcinoma (MRCC) patients (pts) with IL-2 failure in first-line | one year

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of the capecitabine and interferon combination | one year
Evaluate response rate and overall survival with the capecitabine and interferon combination in MRCC pts with progression on IL-2 based regimens | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ilya V. Tsimafeyeu, MD, Principal Investigator — Kidney Cancer Research Bureau; Lev V. Demidov, MD, DSc., Study Director — N.N. Blokhin Russian Cancer Research Bureau
Locations (1):
- N.N. Blokhin Russian Cancer Research Center, Moscow, Russia